CLINICAL TRIAL: NCT06356103
Title: Whey-Based Partially Hydrolyzed Formula Versus Polymeric Formula On Undernourished Neurologically Impaired Children: Open-labelled Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0107060
Record Dates: First submitted 2024-03-16; First posted 2024-04-10 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2022-02

CONDITIONS: Nutrition Disorder, Child; Neurologic Disorder
Keywords: Neurological Impairment; Children; Partially Hydrolyzed Formula
MeSH Terms: conditions — Child Nutrition Disorders; Nervous System Diseases; Neurologic Manifestations

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): received 50% of their caloric requirements as isocaloric polymeric formula (standard ) and 50% standard nutritional feeding according to ESPGHAN guidelines
  Interventions: Dietary Supplement: received 50% of their caloric requirements as isocaloric polymeric formula (standard ) and 50% standard nutritional feeding according to ESPGHAN guidelines
- Group II (Active Comparator): received 50% of their caloric requirements as WPHF and the other 50% as standard nutritional feeding
  Interventions: Dietary Supplement: Whey-Based Partially Hydrolyzed Formula

INTERVENTIONS:
Dietary Supplement: Whey-Based Partially Hydrolyzed Formula — Peptamen junior, 100 kcal/100 ml (Nestlé Health Science, Vevey, Switzerland).
  Arms: Group II
Dietary Supplement: received 50% of their caloric requirements as isocaloric polymeric formula (standard ) and 50% standard nutritional feeding according to ESPGHAN guidelines — protein and micronutrient requirements according to the recommended dietary allowance (RDA)
  Arms: Group I

SUMMARY:
Purpose: Undernutrition is common in neurologically impaired children. It increases the burden of comorbidities and affects the quality of life of these children. This study aimed primarily to compare the efficacy of whey-based partially hydrolyzed formula (WPHF) versus isocaloric polymeric formula on the nutritional status reflected by growth parameters and feeding tolerance in undernourished children with neurological impairment (NI). The secondary aim was to follow up on the changes in these parameters after using WPHF for 3 and 6 months

DETAILED DESCRIPTION:
This prospective open-label randomized study was conducted over 6 months on children with NI aged 2- 6 years. Patients were divided into two groups: one group received 50% of their caloric requirements as isocaloric polymeric formula (standard ) and 50% standard nutritional feeding according to ESPGHAN guidelines (group I), the second group received 50% of their caloric requirements as WPHF, and the other 50% standard nutritional feeding according to ESPGHAN guidelines (group II). At the start of the study, detailed clinical and nutritional history was recorded for all children in the two groups. Anthropometric measurements were measured, and the Z score was calculated for all parameters. Symptoms of feeding intolerance and frequency of chest infections were assessed and reported. These parameters were reassessed after 3 months and 6 months of nutritional intervention and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged from 2-6 years
2. undernourished children with NI (1 or more of the following signs for identification of undernutrition in the studied children:

   * weight for age z score <-2,
   * triceps skinfold thickness <10th centile for age,
   * mid-upper arm fat or muscle area <10th percentile for age,
   * faltering weight
   * failure to thrive.
   * physical signs of undernutrition such as decubitus skin problems and poor peripheral circulation

Exclusion Criteria:

* NI due to metabolic diseases

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of whey-based partially hydrolyzed formula versus standard feeding on the weight in kilogram in undernourished children with neurological impairment (NI). | 6 months
  Identify the Efficacy Of Whey-Based Partially Hydrolyzed Formula on the weight in Kilogram measured using the double weighing method (weight of the parent subtracted from the combined weight of parent and child) on a digital scale.
To compare the efficacy of whey-based partially hydrolyzed formula versus standard feeding on the height/length in centimeter in undernourished children with neurological impairment (NI). | 6 months
  Identify the Efficacy Of Whey-Based Partially Hydrolyzed Formula on the height/length in Centimeter measured by a stadiometer. In children with joint contractions, spasticity, and/or scoliosis, the length was measured by segmental length measurements using sliding calipers. Then the length was estimated by simple equations such as knee-heel length (L = (2.69 x KH) + 24.2), tibia length (L = (3.26 x TL) + 30.8).
To compare the efficacy of whey-based partially hydrolyzed formula versus standard feeding on the body mass index (BMI) in children with neurological impairment (NI). | 6 months
  Identify the Efficacy Of Whey-Based Partially Hydrolyzed Formula on the body mass index (BMI) calculated as [weight in kg]/ [height in m]2
To compare the efficacy of whey-based partially hydrolyzed formula versus standard feeding on the head circumference in centimeter in undernourished children with neurological impairment (NI) | 6 months
  Identify the Efficacy Of Whey-Based Partially Hydrolyzed Formula on the head circumference (HC) in Centimeter measured by non-stretchable tape

SECONDARY OUTCOMES:
To follow up the efficacy of whey-based partially hydrolyzed formula versus standard feeding on the weight in kilogram in undernourished children with neurological impairment (NI) for 3 and 6 months | 6 months
  Follow up the Efficacy Of Whey-Based Partially Hydrolyzed Formula on the weight in Kilogram measured using the double weighing method (weight of the parent subtracted from the combined weight of parent and child) on a digital scale for 3 and 6 months
To follow up the efficacy of whey-based partially hydrolyzed formula versus standard feeding on the height/length in Centimeter in undernourished children with neurological impairment (NI) for 3 and 6 months | 6 months
  Follow up the Efficacy Of Whey-Based Partially Hydrolyzed Formula on the height/length in Centimeter measured by a stadiometer. In children with joint contractions, spasticity, and/or scoliosis, the length was measured by segmental length measurements using sliding calipers. Then, the length was estimated by simple equations such as knee-heel length (L = (2.69 x KH) + 24.2), tibia length (L = (3.26 x TL) + 30.8) for 3 and 6 months.
To follow up the efficacy of whey-based partially hydrolyzed formula versus on the body mass index in undernourished children with neurological impairment (NI) for 3 and 6 months | 6 months
  Follow up the Efficacy Of Whey-Based Partially Hydrolyzed Formula on the body mass index (BMI) calculated as [weight in kg]/ [height in m]2 for 3 and 6 months
To follow up the efficacy of whey-based partially hydrolyzed formula versus standard feeding on the head circumference in Centimeter in undernourished children with neurological impairment (NI) for 3 and 6 months | 6 months
  Follow up the Efficacy Of Whey-Based Partially Hydrolyzed Formula on the head circumference (HC) in Centimeter measured by non-stretchable tape for 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Children Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No